CLINICAL TRIAL: NCT05798403
Title: Electroacupuncture Versus Solifenacin Succinate for Female Overactive Bladder: A Multicenter, Randomized, Controlled, Noninferiority Trial
Brief Title: Efficacy of Electroacupuncture Versus Solifenacin Succinate for Female Overactive Bladder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yin Ping (Other)
Collaborators: Longhua Hospital (Other)
Responsible Party: Sponsor-Investigator, Yin Ping, Shanghai University of Traditional Chinese Medicine, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHDC12022103
Record Dates: First submitted 2023-03-10; First posted 2023-04-04 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Electroacupuncture; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: During the study, except for acupuncturists, other people involved in the trial, including participants, study supervisors, efficacy evaluators, data analysts, prescription drug prescribers and statistical analysts, will all be blinded to patients group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electroacupuncture group (Experimental): Participants will receive electroacupuncture treatment at Shenshu (BL23), Ciliao (BL32), Zhonglvshu (BL29), Huiyang (BL35), Weizhong (BL40), Zhongji (CV3), Dahe (KI12), Shuidao (ST28), Sanyinjiao (SP6). It should be noted that CV3, KI12, ST28, SP6 are used as the group A acupoints and BL23, BL32, BL29, BL35, BL40 as the group B acupoints. Patients will be treated with alternating group A and B acupoints. The frequency of treatment is 3 times a week and each treatment will last for 30 minutes for a total of 12 sessions over the course of four weeks. The follow-up observation will be recorded on week 8 and 16.
  At the same time, participants will also receive placebo medication. Oral Solifenacin Succinate placebo will be used and taken once a day for 4 weeks.
  Interventions: Device: electroacupuncture
- Solifenacin Succinate group (Active Comparator): Participants will take Solifenacin Succinate (Wuhan Human well Puracap (Likang) Pharmaceuticals Co., Ltd.) orally before breakfast for 4 consecutive weeks at 5 mg (1 tablet) per day.
  At the same time, the participants will receive sham electroacupuncture with a pragmatic placebo needle on sham acupoints. Participants will have the same needle retention time, treatment time, and follow-up time as the electroacupuncture group.
  Interventions: Drug: Solifenacin Succinate Tablets

INTERVENTIONS:
Device: electroacupuncture — All acupuncture locations will be sterilized on a routine basis. As acupuncture needles are inserted, all needles will be lifting, twirling, and thrusting to reach de qi, a sensation generally associated with acupuncture, including swelling, soreness, numbness, and heaviness.
  An electrical stimulator is applied to ipsilateral BL32 and BL35 (KI12 and ST28) with continuous waves of 30 Hz and currents of 1 to 5.0 mA. During the study, oral Solifenacin Succinate placebo will be used.
  Other Names: placebo medication
  Arms: Electroacupuncture group
Drug: Solifenacin Succinate Tablets — During the study, participants will take Solifenacin Succinate. The acupuncture points are the same as the electroacupuncture group, without the insertion of needles. The procedures, electrode positions and other treatment settings are the same as the electroacupuncture group, without the skin penetration, power output or needle manipulation of the de qi. At the end of the treatment, the acupuncturist will press the acupuncture point with a dry cotton ball to allow the patient to feel the "needles"being pulled out.
  Other Names: Sham electroacupuncture
  Arms: Solifenacin Succinate group

SUMMARY:
Through a scientific and standardized multicenter, blinding, double-dummy, randomized controlled, noninferiority clinical trial study method, the investigators evaluated electroacupuncture as a safe and effective non-pharmacological treatment for OAB in women by comparison with Solifenacin Succinate.

DETAILED DESCRIPTION:
Epidemiological researches have shown that approximately 500 million people worldwide are affected by OAB, 2 3 with a higher incidence in women than that in men. Pharmacological treatment remains the usual method of clinical treatment. However, some Pharmacologphy has certain side effects, such as blurred consciousness, dry mouth, constipation, and so on, which have limited its widespread clinical use. Therefore, the treatment of OAB needs comprehensive consideration in clinical practice, which deserves our attention and active exploration of other effective treatment methods to relieve patients' pain.Electroacupuncture can effectively improve the clinical symptoms of OAB. As for the comparison between electroacupuncture and medication for the treatment of OAB in women, the results are inconclusive based on the limited research evidence. The aim of the study is to investigate the effectiveness and safety of electroacupuncture compared to Solifenacin Succinate.

ELIGIBILITY:
Inclusion Criteria:

* Meet the American Urological Association (AUA) diagnostic criteria for adult overactive bladder disorder (non-neurogenic) and the Chinese Urological Association's Guidelines for the Diagnosis and Treatment of Urological Diseases in China (2014 edition) for OAB.
* Female patients aged 18-75 years.
* Duration of illness with OAB ≥ 3 months.
* 3≤OABSS≤11.
* No abnormality in routine urine tests.
* Patients had never received acupuncture treatment.
* No mental or intellectual abnormalities, able to understand the provisions of the scales and complete the assessment.
* Consent to participate in this study and sign a written informed consent.

Exclusion Criteria:

* Combination of more serious heart, liver, kidney and other serious diseases; Or patients with severe liver or kidney insufficiency.
* Patients with pelvic organ prolapse ≥ Ⅱ degree, urinary system surgery history or pelvic floor surgery history.
* Patients with other diseases presenting with OAB symptoms.
* Those with urinary diseases (such as calculi and tuberculosis of the bladder), malignant tumors, and neurological disorders.
* Patients who are pregnant or breastfeeding.
* Patients using medication that may affect bladder function one month prior to enrollment or having received behavioural therapy for OAB three months prior to enrolment, etc.
* Patients with pacemakers.
* Patients with blood diseases, diabetes mellitus or mental diseases.
* Infections, ulcers, abscesses, and skin infections at needling sites; metal allergy or extreme needle phobia.
* Participation in other clinical medical trial studies over the last month.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
the percentage change in the number of voids every 24 hours at week 4. | At week 4 (end of treatment).
  The percentage change in the number of voids every 24 hours at week 4 compared to baseline. It is measured by a three-day voiding diary.

SECONDARY OUTCOMES:
The percentage change in the number of voids every 24 hours. | At week 2, week 8(follow-up) and week 16 (follow-up).
  The percentage change in the number of voids every 24 hours at 2th, 8th and 16th weeks of the trail.It is measured by a three-day voiding diary.
The mean changes of OABSS. | At week 2, 4 (end of treatment), week 8(follow-up) and week 16 (follow-up).
  The OABSS assessed the occurrence of daytime voiding, nocturnal voiding, urgency and urge incontinence in patients during the last week.
The number of urinary incontinence and urgency every 24 hours. | At week 2, 4 (end of treatment), week 8(follow-up) and week 16 (follow-up).
  The number of urinary incontinence and urgency every 24 hours based on a three-day voiding diary.
Overactive Bladder Questionnaire (OAB-q). | At baseline and week 4 (end of treatment).
  The OAB-q is an observation of the severity and frequency of bladder-related symptoms in patients over the past four weeks.
Generalized Anxiety Disorder 7 (GAD-7) | At baseline and week 4 (end of treatment).
  The GAD-7 is used to assess subjects' anxiety.
Health-Related Quality of Life (HRQoL) | At baseline and week 4 (end of treatment).
  The HRQoL will be measured by the King's Health Questionnaire (KHQ).
Participants'self-evaluation of therapeutic effects. | At week 2, 4 (end of treatment), week 8(follow-up) and week 16 (follow-up).
  It will be evaluated using a four-point scale, which is level 0 (not at all helpful), level 1 (a little helpful), level 2 (moderately helpful) and level 3 (very helpful).

OTHER OUTCOMES:
Incidence of adverse events | During 1-4 weeks.
  Observe the incidence of adverse events during the treatment.
Evaluation of discomfort during treatment. | Within 5 minutes after the first, sixth and twelfth acupuncture treatment.
  Visual analog scale (VAS) will be used to evaluate the degree of discomfort during treatment. The scale ranging from 0 to 10cm, with 0cm indicating no discomfort and 10cm indicating severe discomfort. Evaluation time: The average value of the first and ninth acupuncture treatments was taken within 5 minutes after the end of the two treatments. If the VAS value is missing in one of the cases, another is taken as the result.
Patient acceptability evaluation | Within 5 minutes after the first and ninth acupuncture treatment.
  0=very difficult to accept, 1=slightly difficult to accept, 2=acceptable, 3=easy to accept, 4=very easy to accept. Evaluation time: The average value of the first and ninth acupuncture treatments was taken within 5 minutes after the end of the two treatments. If the VAS value is missing in one of the cases, another is taken as the result.
Blinding assessment | At the end of the 12th session of acupuncture treatment
  Six options will be offered by an independent assessor in an interrogative manner: electroacupuncture, sham electroacupuncture and indeterminate; medication, placebo treatment and indeterminate. The patients' answers will be statistically analyzed to assess the success of the blinded implementation.

CONTACTS AND LOCATIONS:
Overall Officials: YUELAI CHEN, Principal Investigator — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Longhua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lightner DJ, Gomelsky A, Souter L, Vasavada SP. Diagnosis and Treatment of Overactive Bladder (Non-Neurogenic) in Adults: AUA/SUFU Guideline Amendment 2019. J Urol. 2019 Sep;202(3):558-563. doi: 10.1097/JU.0000000000000309. Epub 2019 Aug 8. PMID 31039103
- [Background] Joseph S, Maria SA, Peedicayil J. Drugs Currently Undergoing Preclinical or Clinical Trials for the Treatment of Overactive Bladder: A Review. Curr Ther Res Clin Exp. 2022 Apr 6;96:100669. doi: 10.1016/j.curtheres.2022.100669. eCollection 2022. PMID 35494662
- [Background] Mirzaei M, Daneshpajooh A, Anvari SO, Dozchizadeh S, Teimorian M. Evaluation of the Clinical Efficacy and Complications of Duloxetine in Comparison to Solifenacin in the Treatment of Overactive Bladder Disease in Women: A Randomized Clinical Trial. Urol J. 2021 Aug 3;18(5):543-548. doi: 10.22037/uj.v18i.6274. PMID 34346046
- [Background] Hargreaves E, Harding C, Clarkson C. Acupuncture in addition to standard conservative treatment for overactive bladder; a feasibility trial for a randomized controlled study. Neurourol Urodyn. 2021 Sep;40(7):1770-1779. doi: 10.1002/nau.24741. Epub 2021 Jul 21. PMID 34289514
- [Derived] Chen B, Yin P, Li J, Hou W, Fan Q, Huai Y, Liu L, Hu J, Chow ST, Li X, Ming S, Chen YL. Electroacupuncture versus solifenacin succinate for female overactive bladder: study protocol for a multicentre, randomised, controlled, double-dummy, non-inferiority trial. BMJ Open. 2024 Sep 12;14(9):e076374. doi: 10.1136/bmjopen-2023-076374. PMID 39266323